CLINICAL TRIAL: NCT06919445
Title: Novel Mobile Resource for Food Insecurity Randomized Controlled Trial
Brief Title: Novel Mobile Resource for Food Insecurity
Acronym: NO MORE FI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cristin Fritz, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 241490
Record Dates: First submitted 2025-03-21; First posted 2025-04-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Food Insecurity
Keywords: mHealth; Pediatric; Food Insecurity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Food Resources Control (No Intervention): Caregivers included in the usual care group receive a paper food resource handout as part of their discharge paperwork. This paper is given to the family and reviewed by the nurse completing their discharge. Families may also meet with a resource navigator during admission if they indicate a desire to talk with someone about food resources during their hospitalization. Finally, all caregivers with FI identified during screening are eligible to receive a food box or frozen meal at the time of discharge from the hospital.
- Usual Food Resources PLUS Text Connect Intervention (Experimental): Caregivers included in the intervention arm receive a 'Text Connect' message with food resource information one day and four days after discharge in addition to the usual care information received by the control group
  Interventions: Other: 'Text Connect' text messages

INTERVENTIONS:
Other: 'Text Connect' text messages — The Text Connect message includes 1) a link to a FindHelp (an online social resource database available in over 100 languages) search tailored to the recipient's home ZIP code 2) information regarding applying for the Supplemental Nutrition Assistance Program (SNAP), and information regarding applying for the Special Supplemental Program for Women, Infants, and Children (WIC). All text message content was initially developed in consultation with caregivers of children with FI identified during an admission through a Community Engagement studio and was approved by the institution's Effective Health Communication Core. The investigators have adapted the content based on feedback from participants in the pilot study.
  Arms: Usual Food Resources PLUS Text Connect Intervention

SUMMARY:
The goal of this clinical trial is to learn if a novel text-message-based intervention is a more effective method for providing food resource information to families of recently hospitalized children who are experiencing food insecurity compared to the current standard practice of a paper handout delivered at the time of hospital discharge. The hypotheses the investigators seek to prove are:

1. That the Text Connect intervention will have greater reach and engagement and be more effective in facilitating connection to food resources than receiving a paper handout alone.
2. That the Text Connect intervention will improve household food security to a greater degree than a paper handout alone.

DETAILED DESCRIPTION:
The mHealth intervention, Text Connect, leverages universal FI screening embedded in the routine clinical care of hospitalized children and offers an innovative approach to providing food resource information that addresses previously identified challenges. The anonymous nature of the text message may empower families with concerns related to sharing their need to pursue resources. Leveraging an already existing online social resource database that is frequently updated and searchable by ZIP Code in many different languages ensures that community program information is accurate, relevant, and tailored to the user's needs. Automated delivery to a personal device addresses the barrier of not receiving referral information and enables patients and families to utilize the information when most convenient for them. Importantly, it is also a promising approach to disseminating this information to all individuals with FI. While development of an app or link in an online portal is a possible electronic information dissemination approach, there are known challenges in accessing such tools that would limit use by many in the population that most frequently experiences FI.

By leveraging an electronic health record vendor's (Epic) native screening questions to identify eligible families and an external social resource database to provide tailored resources, this approach is scalable to other care settings, other domains of needs, and other institutions. Most importantly, successful implementation of this intervention holds the potential to improve family food security and child health outcomes.

The investigator's pilot study testing the feasibility, usability, and acceptability of this proposed approach to resource provision demonstrated that the intervention reaches the majority of the intended population, over half of recipients engage with the content, has excellent usability, and is acceptable to families. Thus, the overarching goal of this proposal is to rigorously test this approach to resource information delivery through a randomized controlled trial to inform health-system approaches to providing social resource information in response to screening. The specific aims are:

Aim 1: In a randomized controlled trial, the investigators will test the reach, engagement, and effectiveness of resource connection of the mHealth intervention, Text Connect, as compared to usual care, a paper resource handout, among families with FI. The investigators hypothesize that the mHealth intervention Text Connect will have greater reach and engagement and be more effective in facilitating connection to food resources than receiving a paper handout alone.

Aim 2: Assess the impact of the Text Connect intervention on household food and nutrition security status, perceived stigma, and trust in the healthcare team compared to usual care. The investigators hypothesize that the Text Connect intervention will improve household food security to a greater degree than a paper handout alone.

ELIGIBILITY:
Inclusion Criteria:

* Must be a caregiver of a child admitted to the hospital
* Must have a positive screening for Food Insecurity documented in the Electronic Health Record as conducted as part of the child's routine clinical care

Exclusion Criteria:

* Primary language other than English or Spanish
* Repeat admission during the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Resource Connection (Effectiveness) | Days 5, 12, and 30
  Effectiveness is measured as the proportion of caregivers who report (Yes/No) getting a new food resource since getting home from their child's hospitalization.
Caregiver-reported Engagement with information | Days 5, 12, and 30
  Measured among control and intervention groups as the proportion of caregivers who report reading (Yes/No) or using the content of the discharge resource handout (control) or text message (intervention) to search for a new resource
System-collected Engagement with information | Days 1 and 4
  Measured among the intervention group as the proportion of caregivers who click on the embedded FindHelp search link
Caregiver-reported Reach | 5, 12, & 30
  Reach will be measured among intervention and control groups as the proportion of caregivers who report receiving the text message (intervention) or paper handout (control)
System-collected Reach | Day 1 and 4
  Will be measured among among the intervention cohort as the proportion of caregivers who have successful delivery of at least one Text Connect intervention message as recorded by Twilio report of text message delivery

SECONDARY OUTCOMES:
Food Security | Day 30
  Food Security is measured by the 18 item USDA Food Security Survey. The items ask about households ability to afford enough food. Raw scores range from 0-18, which are then classified into categories including very low food security (8-18), low food security (3-7), marginal food security (1-2) and high food security (0)
Nutrition Security | Day 30
  Nutrition Security is measured by 4-item Center for Nutrition and Health Impact Nutrition Security Scale. The items ask about caregivers ability to access nutritious foods. Answer choices include 'Never, Rarely, Sometimes, Often, Always, and Don't Know'. Scores range from 0-4, where higher scores indicate higher nutrition
Resilience | Day 30
  Resilience is measured by Center for Nutrition and Health Impact Adaptive Capacity 2-item Screener. The items ask about caregivers ability to find assistance in the face of financial challenges. Answer choices include a 6-point Likert Scale from Strongly Agree to Strongly Disagree, with responses of Slightly Disagree, Disagree, or Strongly Disagree to either question indicating a positive screen for needing additional support to navigate financial challenges.
Stigma | Day 30
  Stigma is measured by a modified version of the Discrimination in Medical Settings scale asking about the child's recent hospitalization. The items ask about negative experiences in the health care setting. Each question is rated on a 5-point Likert scale (1-never, 2-rarely, 3-sometimes, 4-most of the time, 5-always). Scores range from 5-35 with higher scores indicating more experiences of discrimination.
Trust in Health Care System | Day 30
  Trust in health care team is measured by 5-point Likert scale, where higher score indicates higher level of trust.

CONTACTS AND LOCATIONS:
Locations (1):
- Monroe Carell Jr Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No